CLINICAL TRIAL: NCT00985972
Title: Physical Activity and Nutritional Education as School-based Interventions to Control Overweight in Children and Adolescents: a Systematic Review (Project PANE)
Brief Title: Physical Activity and Nutritional Education as School-based Interventions to Control Obesity in Children and Adolescents
Acronym: PANE
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Paulo Henrique de Araujo Guerra, DSc., University of Sao Paulo General Hospital
Other Study IDs: PANE0575-08
Record Dates: First submitted 2009-09-23; First posted 2009-09-29 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: OVERWEIGHT; OBESITY
Keywords: PHYSICAL ACTIVITY; SCHOOL; NUTRITION; EDUCATION; OVERWEIGHT
MeSH Terms: conditions — Overweight; Obesity; Motor Activity | interventions — Exercise; Nutrition Assessment

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Intervention: Groups of school intervention that involves a combination of the physical activity and nutrition education in subjects 6 to 18 years of age
  Interventions: Behavioral: Physical Activity and Nutrition Education
- Control: Groups included in the same school communities that serve as reference for individuals involved in intervention.
  Interventions: Behavioral: Physical Activity and Nutrition Education

INTERVENTIONS:
Behavioral: Physical Activity and Nutrition Education — School-based interventions involving Physical Activity or/and Nutrition Education.

SUMMARY:
The aim of this study focuses on obtaining accurate information on the effectiveness of interventions involving physical activity and/or nutrition education developed in the school environment. This study is intended to assist in future assembly and development of effective school practices related to preventing and reducing levels of overweight in children and adolescents.

Updated data from the systematic review:

5,899 studies were retrieved in 14 databases (Assia, Central Cochrane, CINAHL, EMBASE, ERIC, ISI, LILACS, Physical Education Index, PsycINFO, PubMed, Social Care Online, Social Services Abstracts, Sociological Abstracts, SPORTDiscus)

1,228 were excluded as duplicates by Eppi Reviewer

4,678 studies referred for evaluation by title and abstracts (4,671 by systematic searches, 7 by cross-references list)

211 full text papers reviewed by EPHPP and GRADE tools

140 studies with data extracted

Body Mass Index Results:

1. Guerra PH, Nobre MRC, Silveira JAC, Taddei JAAC. The effect of school-based physical activity interventions on body mass index: a meta-analysis of randomized trials. Clinics (Sao Paulo). 2013 Sep;68(9):1263-1273 - Isolated Physical Activity interventions: 0.02 (95%CI: -0.13, 0.17; 11 trials; n=4,273; I2=77%)
2. Silveira JA, Taddei JA, Guerra PH, Nobre MR. The effect of participation in school-based nutrition education interventions on body mass index: a meta-analysis of randomized controlled community trials. Prev Med. 2013 Mar;56(3-4):237-43 - Isolated Nutrition Education interventions: -0.33 (95%CI: -0.55, -0.11; 8 trials; n=8,491; I2=95%)
3. Guerra PH, Nobre MRC, Silveira JAC, Taddei JAAC. School-based physical activity and nutritional education interventions on body mass index: a meta-analysis of randomized community trials - Project PANE (manuscript under review) - Combined Physical Activity and Nutrition Education interventions: -0.03 (-0.09, 0.04; 38 trials; n=28,870; I2=83%) / All interventions included: -0.03 (95%CI: -0.09, 0.03; 55 trials n=41,634; I2=87%)

DETAILED DESCRIPTION:
The inordinate increase in the prevalence of overweight and obesity at the international level today is one of the targets of concern the department of public health, and gradually has been the focus of many studies and interventions which emphasize the need for more evidence to clear and effective its prevention and reduction. Obesity can affect the short or long term health of individuals, through problems such as left ventricular hypertrophy in young-adult and atherosclerosis, which is due to the formation of plaques of fat in the arterial wall and may lead to coronary artery disease , cerebrovascular disease and peripheral vascular disease.

The promotion of regular practice of physical activity through physical education school can be an effective way to prevent obesity among children, especially girls. There is an inverse relationship between physical activity and incidence of hypertension. The earlier the entrance to the practice of physical activities, there will be more effective in combating the increase in body mass index (BMI).

Nutrition Education is to extend the knowledge on nutrition and the ability to understand the practices and eating behavior, improving the relationship of the individual in the environment which is introduced, allowing the taking of decisions under the situation presented.

ELIGIBILITY:
Inclusion Criteria:

* Randomized clinical / community trials whose main objective is the focus on control and / or reduction of body weight of the participants, conducted by a program developed in the scholar environment that promotes the practice of physical activity and healthy eating through nutrition education.
* Studies that include participants aged 6 to 18 years of age, regardless of the range of weight.
* There is no restriction ethnic, social, gender, nutritional status and physical fitness.
* There is no limitation of language for critical evaluation of studies.

Exclusion Criteria:

* Studies making use of pharmacological agents
* Studies with participants who suffer from diseases, or specific clinical conditions, except obesity
* Studies not conducted in the school environment
* The duplicated data will be excluded.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children and adolescents aged 6 to 18 years of age included in the school environment, regardless of their ethnicity, social condition and weight range.
Sampling Method: Probability Sample
Enrollment: 41634 (Actual)
Dates: Start 2009-06; Primary Completion 2010-12 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | Assessments results should at least monitor the execution time of the intervention studies, with a minimum of two assessments: pre-and post-intervention. This requirement depends directly on the studies to be extracted in the systematic search.

SECONDARY OUTCOMES:
Body Weight | requirement for pre and post-intervention assessments
Blood Pressure | requirement for pre and post-intervention assessments
  Systolic and Diastolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Moacyr MR Nobre, PhD, Principal Investigator — University of São Paulo, Faculty of Medicine, Heart Institute (InCor), Clinical Epidemiology Unit; Paulo Henrique A Guerra, DSc, Principal Investigator — University of São Paulo, Faculty of Medicine, Heart Institute (InCor), Clinical Epidemiology Unit; Jonas A Silveira, MSc, Principal Investigator — Federal University of São Paulo, Department of Pediatrics
Locations (1):
- Heart Institute, General Hospital of Faculty of Medicine of University of Sao Paulo (InCor HCFMUSP), São Paulo, São Paulo, Brazil

REFERENCES:
- [Result] Silveira JA, Taddei JA, Guerra PH, Nobre MR. Effectiveness of school-based nutrition education interventions to prevent and reduce excessive weight gain in children and adolescents: a systematic review. J Pediatr (Rio J). 2011 Sep-Oct;87(5):382-92. doi: 10.2223/JPED.2123. English, Portuguese. PMID 22012577
- [Result] Silveira JA, Taddei JA, Guerra PH, Nobre MR. The effect of participation in school-based nutrition education interventions on body mass index: a meta-analysis of randomized controlled community trials. Prev Med. 2013 Mar;56(3-4):237-43. doi: 10.1016/j.ypmed.2013.01.011. Epub 2013 Jan 29. PMID 23370048
- [Result] Guerra PH, Nobre MR, Silveira JA, Taddei JA. The effect of school-based physical activity interventions on body mass index: a meta-analysis of randomized trials. Clinics (Sao Paulo). 2013 Sep;68(9):1263-73. doi: 10.6061/clinics/2013(09)14. PMID 24141844
- [Result] Guerra PH, Nobre MR, da Silveira JA, Taddei JA. School-based physical activity and nutritional education interventions on body mass index: a meta-analysis of randomised community trials - project PANE. Prev Med. 2014 Apr;61:81-9. doi: 10.1016/j.ypmed.2014.01.005. Epub 2014 Jan 16. PMID 24440161